CLINICAL TRIAL: NCT04313192
Title: Optimal Frequency Used in Transcutaneous Electrical Nerve Stimulation (TENS) for Treating Nocturnal Enuresis in Children
Brief Title: TENS Treatment for Bedwetting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Adam Howe, MD, Assistant Professor of Surgery, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5618
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Nocturnal Enuresis; Bed Wetting
Keywords: Nocturnal Enuresis; Bedwetting; TENS
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Pulse rate 2Hz (hertz) (Experimental): electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 2 Hz, intensity setting to patient's tolerance, duration 30 days
  Interventions: Device: pulse rate of 2 Hz
- Pulse rate 10Hz (Experimental): electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 10 Hz, intensity setting to patient's tolerance, duration 30 days
  Interventions: Device: pulse rate of 10 Hz
- Pulse rate 150Hz (Experimental): electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 150 Hz, intensity setting to patient's tolerance, duration 30 days
  Interventions: Device: pulse rate of 150 Hz

INTERVENTIONS:
Device: pulse rate of 2 Hz — electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 2 Hz, intensity setting to patient's tolerance, duration 30 days
  Other Names: TENS
  Arms: Pulse rate 2Hz (hertz)
Device: pulse rate of 10 Hz — electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 10 Hz, intensity setting to patient's tolerance, duration 30 days
  Other Names: TENS
  Arms: Pulse rate 10Hz
Device: pulse rate of 150 Hz — electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 150 Hz, intensity setting to patient's tolerance, duration 30 days
  Other Names: TENS
  Arms: Pulse rate 150Hz

SUMMARY:
Children referred to pediatric urology clinic for primary nocturnal enuresis will be screened for enrollment. Patients who fail will next be offered therapy with a bedwetting alarm device or a TENS unit as an alternative, and those who chose TENS therapy will be included in the study.The patients will be randomized into three groups of 30 patients each. Group 1 will be the long frequency set at 2 Hz (hertz). Group 2 will be the moderate frequency set at 10 Hz. Group 3 will be the short frequency set 150 Hz. The patients will be provided with a TENS unit and electrode pads and caretakers instructed on how to use the apparatus.

The child's TENS unit will be set at a frequency determined by randomization, pulse width of 260 seconds, and an intensity to be determined in the office based upon when the child feels sensitive to the TENS unit. The child will be randomized and will place the electrodes along the posterior tibial nerve on the medial ankle each night before bed time for 15 minutes for a total of 30 days. Diaries including nighttime incontinence episodes and a "wet sheet" scale (dry, damp, wet, soaked) will be recorded, along with any adverse reactions to the TENS unit. Patients will be followed up after one month of TENS with evaluation including the Pediatric Urinary Incontinence Questionnaire, a validated tool for measuring quality of life in children with bladder dysfunction; this questionnaire will be filled out prior to starting TENS treatment in order to compare the effect of treatment on QOL. The data will be collected at different time points (baseline and after 1 month of treatment) for each group by itself and the groups compared against each other using statistical analysis.

DETAILED DESCRIPTION:
Institutional review board approval was obtained. Children ages 5-18 years old referred to the pediatric urology clinic for primary nocturnal enuresis will be screened for enrollment. Behavioral modification (limiting evening drinking, double voiding prior to bedtime, bowel habits, social anxiety factors) will be utilized first. Patients who fail will next be offered therapy with a bedwetting alarm device or a TENS unit as an alternative, and those who chose TENS therapy will be included in the study. Patients who have previously tried pharmacologic treatment for nocturnal enuresis or alternative therapy for urologic disorders within the past 30 days, daytime incontinence symptoms, known "high volume" voiders (determined from history), bedwetting episodes on the average of less than one time per week, medications predisposing to incontinence (eg, Lithium for bipolar disorder), other known voiding or neurologic disorders (eg, overactive bladder, myelomeningocele), secondary etiologies for nocturnal enuresis (eg, cystitis, obstructive sleep apnea, urinary fistulae), prior use of a TENS unit or other neuromodulation for bedwetting, and any contraindications to usage of a TENS unit such as having a pacemaker will be excluded. Patients who have previously tried the bedwetting alarm will not be excluded from the study.

The patients will be randomized into three groups of 30 patients each. Group 1 will be the long frequency set at 2 Hz. Group 2 will be the moderate frequency set at 10 Hz. Group 3 will be the short frequency set 150 Hz. There is no sham group in this study as the investigator has previously found posterior tibial TENS to be effective and lasting, and as such all patients will be treated. The investigator will aim to recruit 30 patients per group for a total of 90 patients. Detailed explanation of the purpose if the study, along with the risks and benefits of TENS will be given to the patient and caretakers by a provider prior to obtaining informed consent for enrollment into the study. The patients will be provided with a TENS unit and electrode pads and caretakers instructed on how to use the apparatus.

Parents/patients of enrolled patients will fill out nightly voiding diaries, recording nighttime incontinence episodes and subjective "wet sheets" scale per night (dry, damp, wet, soaked) for 30 days prior to randomization into the treatment arms. The TENS sessions will be performed nightly at bedtime for 15 minutes for 30 days. TENS units will be set at a frequency of 10Hz, and intensity determined in the office by the sensitivity threshold of the patient. Voiding diaries will be kept each night while on TENS therapy. A voiding diary will also be completed 30 days before TENS treatment, patients and families will fill out the Pediatric Urinary Incontinence Questionnaire (PIN-Q), a validated tool for measuring quality of life in children with bladder dysfunction. Patients will follow up at day 30 and as needed (worsening symptoms, adverse reactions, concerns, and questions regarding usage of TENS). Patients who record 2 wet nights per week (a total of 8/30=27% wet nights) will be eligible for the TENS study. Those who record less than 2 wet nights per week will be ineligible for the TENS study but will be offered therapy using a bedwetting alarm device or other treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting with nocturnal enuresis (more than 1x a week)
2. Failed Behavioral modification treatment (limiting evening drinking, double voiding prior to bedtime, bowel habits, social anxiety factors)
3. Ability to provide informed consent and assent and complete study requirements

Exclusion Criteria:

1. Patients who have previously tried pharmacologic treatment for nocturnal enuresis, neuromodulation or other alternative therapy for urologic disorders within the past 30 days
2. Daytime incontinence symptoms
3. Known "high volume" voiders (determined from history)
4. Bedwetting episodes on the average of less than two times per week,
5. Medications predisposing to incontinence (eg, Lithium for bipolar disorder)
6. Other known voiding or neurologic disorders (eg, overactive bladder, myelomeningocele, interstitial cystitis, etc)
7. Secondary etiologies for nocturnal enuresis (eg, cystitis, obstructive sleep apnea, urinary fistulae, heart disease)
8. Any contraindications to usage of a TENS unit (pacemaker or other implantable device, lymphedema, pregnancy, malignancy,bleeding or clotting disorders, unhealthy tissue, seizure disorders, impaired cognition)
9. Any history of heart disease or complications

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of wet nights | 30 days
  Total number of change in wet nights compared in each TENS arm and baseline wet nights

SECONDARY OUTCOMES:
Severity of wet nights | 30 days
  Mean score (0 dry to 3 soaked) of subjective severity of wetness each night during treatment month compared to baseline month
Pediatric Incontinence Questionnaire (PIN-Q) | 30 days
  Quality of life questionnaire score after treatment month compared to after baseline month. Scores = mild <20, moderate 21-50, and severe >51

CONTACTS AND LOCATIONS:
Overall Officials: Adam Howe, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States

REFERENCES:
- [Background] Alcantara AC, Mello MJ, Costa e Silva EJ, Silva BB, Ribeiro Neto JP. Transcutaneous electrical neural stimulation for the treatment of urinary urgency or urge-incontinence in children and adolescents: a Phase II clinica. J Bras Nefrol. 2015 Jul-Sep;37(3):422-6. doi: 10.5935/0101-2800.20150065. English, Portuguese. PMID 26398655
- [Background] Barroso U Jr, Lordelo P, Lopes AA, Andrade J, Macedo A Jr, Ortiz V. Nonpharmacological treatment of lower urinary tract dysfunction using biofeedback and transcutaneous electrical stimulation: a pilot study. BJU Int. 2006 Jul;98(1):166-71. doi: 10.1111/j.1464-410X.2006.06264.x. PMID 16831163
- [Background] Barroso U Jr, Viterbo W, Bittencourt J, Farias T, Lordelo P. Posterior tibial nerve stimulation vs parasacral transcutaneous neuromodulation for overactive bladder in children. J Urol. 2013 Aug;190(2):673-7. doi: 10.1016/j.juro.2013.02.034. Epub 2013 Feb 16. PMID 23422257
- [Background] Bjorkstrom G, Hellstrom AL, Andersson S. Electro-acupuncture in the treatment of children with monosymptomatic nocturnal enuresis. Scand J Urol Nephrol. 2000 Feb;34(1):21-6. doi: 10.1080/003655900750016832. PMID 10757265
- [Background] Bouali O, Even L, Mouttalib S, Moscovici J, Galinier P, Game X. [Tibial nerve transcutaneous stimulation for refractory idiopathic overactive bladder in children and adolescents]. Prog Urol. 2015 Sep;25(11):665-72. doi: 10.1016/j.purol.2015.04.005. Epub 2015 May 26. French. PMID 26022237
- [Background] Bower WF, Wong EMC, Yeung CK. Development of a validated quality of life tool specific to children with bladder dysfunction. Neurourol Urodyn. 2006;25(3):221-227. doi: 10.1002/nau.20171. PMID 16496391
- [Background] Chen ML, Chermansky CJ, Shen B, Roppolo JR, de Groat WC, Tai C. Electrical stimulation of somatic afferent nerves in the foot increases bladder capacity in healthy human subjects. J Urol. 2014 Apr;191(4):1009-13. doi: 10.1016/j.juro.2013.10.024. Epub 2013 Oct 7. PMID 24113017
- [Background] Chen YJ, Zhou GY, Jin JH. [Transcutaneous electrical acupoint stimulation combined with auricular acupoint sticking for treatment of primary nocturnal enuresis]. Zhongguo Zhen Jiu. 2010 May;30(5):371-4. Chinese. PMID 20518171
- [Background] Lordelo P, Benevides I, Kerner EG, Teles A, Lordelo M, Barroso U Jr. Treatment of non-monosymptomatic nocturnal enuresis by transcutaneous parasacral electrical nerve stimulation. J Pediatr Urol. 2010 Oct;6(5):486-9. doi: 10.1016/j.jpurol.2009.11.005. PMID 20837326
- [Background] Lordelo P, Teles A, Veiga ML, Correia LC, Barroso U Jr. Transcutaneous electrical nerve stimulation in children with overactive bladder: a randomized clinical trial. J Urol. 2010 Aug;184(2):683-9. doi: 10.1016/j.juro.2010.03.053. Epub 2010 Jun 18. PMID 20561643
- [Background] de Oliveira LF, de Oliveira DM, da Silva de Paula LI, de Figueiredo AA, de Bessa J Jr, de Sa CA, Bastos Netto JM. Transcutaneous parasacral electrical neural stimulation in children with primary monosymptomatic enuresis: a prospective randomized clinical trial. J Urol. 2013 Oct;190(4):1359-63. doi: 10.1016/j.juro.2013.03.108. Epub 2013 Mar 29. PMID 23545102
- [Background] Tai C, Shen B, Chen M, Wang J, Liu H, Roppolo JR, de Groat WC. Suppression of bladder overactivity by activation of somatic afferent nerves in the foot. BJU Int. 2011 Jan;107(2):303-9. doi: 10.1111/j.1464-410X.2010.09358.x. PMID 20394612
- [Background] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027
- [Background] ELECTROPHYSICAL AGENTS - Contraindications And Precautions: An Evidence-Based Approach To Clinical Decision Making In Physical Therapy. Physiother Can. 2010 Fall;62(5):1-80. doi: 10.3138/ptc.62.5. Epub 2011 Jan 5. No abstract available. PMID 21886384
- [Background] Robertson Val, Ward A, Low J, Reed A. Electrotherapy explained: principles and practice (4th edition). Elsevier Ltd (UK), 2006.
- [Background] Sharma M, Aggarwal V, Bahadur R, Gupta R. Burns secondary to improper usage of transcutaneous electrical nerve stimulation: a case report. Pb J Ortho. 2011;12(1):72-3.
- [Background] Howe et al. Transcutaneous electric nerve stimulation (TENS) for the treatment of nocturnal enuresis in children. [NOT YET IN PRESS]
- [Background] Moeller Joensson I, Hagstroem S, Siggaard C, Bower W, Djurhuus JC, Krogh K. Transcutaneous Electrical Nerve Stimulation Increases Rectal Activity in Children. J Pediatr Gastroenterol Nutr. 2015 Jul;61(1):80-84. doi: 10.1097/MPG.0000000000000802. PMID 25844704